CLINICAL TRIAL: NCT00288912
Title: Self-Management of Osteoarthritis: A Tailored, Telephone-based Intervention
Brief Title: Self-Management of Osteoarthritis
Acronym: SeMOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 04-016
Record Dates: First submitted 2006-02-06; First posted 2006-02-08 (Estimated); Results first posted 2014-09-12 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Osteoarthritis
Keywords: Self-Care; Telemedicine; Pain; Veterans
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Health Education Intervention (Active Comparator): Health Education Intervention
  Interventions: Behavioral: Health Education
- Usual Medical Care (No Intervention): Usual Medical Care
- Osteoarthritis Self-Management (Experimental): Osteoarthritis Self-Management
  Interventions: Behavioral: Osteoarthritis Self-Management

INTERVENTIONS:
Behavioral: Health Education — 12-month intervention consisting of monthly phone calls about common health conditions and screening. Also includes written educational materials on these topics.
  Arms: Health Education Intervention
Behavioral: Osteoarthritis Self-Management — 12-month intervention consisting of monthly phone calls about topics related to self-care for osteoarthritis. Also includes written educational materials on these topics. Participants set goals and action plans, with assistance from health educator, about managing their osteoarthritis.
  Arms: Osteoarthritis Self-Management

SUMMARY:
The purpose of this study is to examine whether a telephone-based self-management intervention improves pain, physical function, and other outcomes among veterans with osteoarthritis of the hip or knee.

DETAILED DESCRIPTION:
Background / Rationale: Osteoarthritis (OA) is the one of the most common chronic conditions among veterans, and over half of VA health care users with OA report being limited in their daily activities because of joint symptoms. However, studies have not examined interventions to improve outcomes or quality of care among the large and growing number of veterans with OA. Telephone-based self-management interventions may be a cost-effective way to improve pain, physical function, and other outcomes in this patient population. Objective: The purpose of this study is to examine the effectiveness of a one-year telephone-based self-management intervention for veterans with hip or knee OA. The primary hypothesis is that the self-management intervention will result in a greater reduction in pain as compared to both usual care and attention control conditions. Methods: This will be a randomized control trial of 519 veterans at the Durham VAMC who have radiographic evidence and a physician diagnosis of OA of the hip or knee. Participants will be equally allocated to self-management, attention control, and usual care groups. The self-management intervention is designed to provide participants with key information about OA and its treatment and to enhance participants' self-efficacy for managing OA-related symptoms. This intervention will involve provision of written, audio, and video educational materials, as well as monthly telephone calls by a nurse. The nurse will guide participants in developing personal OA-related goals, as well as specific plans for meeting these goals. Other strategies for enhancing self-efficacy will include modeling and mastery of self-management behaviors, persuasion to adopt these behaviors, and reinterpretation of OA symptoms. The attention control group will receive written materials on health screening related topics (not OA-related), and the nurse will call participants on a monthly basis to discuss these materials. The primary outcome measure for this study will be self-reported pain (Arthritis Impact Measurement-2 (AIMS2) subscale), and secondary outcomes will be self-reported function (AIMS2 subscale), affect (AIMS2 subscale), and arthritis specific self-efficacy. Outcomes will be measured at baseline and following the one-year study period. Analysis of covariance will be used to compare primary and secondary outcomes between the intervention group and each of the control groups, adjusting for baseline measures, participant demographic and clinical characteristics. We will also examine the cost-effectiveness of the intervention. Impact: This study is significant because it examines a highly prevalent but understudied chronic illness among veterans. In addition, this OA self-management program will contribute to the VA health care system's specific mission to improve pain management through patient education and participation. The proposed self-management intervention will be low-cost and easy to disseminate within the VA health care system. Therefore it may be an important tool for improving outcomes, especially pain, among many veterans with OA.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic evidence of hip or knee osteoarthritis
* Current / persistent joint symptoms (pain, aching, stiffness)

Exclusion Criteria:

* Other rheumatic disease (i.e., rheumatoid arthritis, fibromyalgia)
* Hospitalization for stroke or cardiovascular event within past 3 months
* Metastatic cancer
* Active diagnosis of psychosis
* Terminal illness
* On waiting list for arthroplasty
* Resident of nursing home
* Severely impaired in hearing or speech (participants must be able to respond to phone calls)
* Significant cognitive dysfunction
* No access to a telephone
* Current participation in another interventional study for osteoarthritis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 523 (Actual)
Dates: Start 2006-10; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Dominick Allen, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

REFERENCES:
- [Result] Sperber NR, Allen KD, Devellis BM, Devellis RF, Lewis MA, Callahan LF. Differences in effectiveness of the active living every day program for older adults with arthritis. J Aging Phys Act. 2013 Oct;21(4):387-401. doi: 10.1123/japa.21.4.387. Epub 2012 Nov 19. PMID 23170757
- [Result] Sperber NR, Bosworth HB, Coffman CJ, Juntilla KA, Lindquist JH, Oddone EZ, Walker TA, Weinberger M, Allen KD. Participant evaluation of a telephone-based osteoarthritis self-management program, 2006-2009. Prev Chronic Dis. 2012;9:E73. Epub 2012 Mar 22. PMID 22440547
- [Result] Sperber NR, Bosworth HB, Coffman CJ, Lindquist JH, Oddone EZ, Weinberger M, Allen KD. Differences in osteoarthritis self-management support intervention outcomes according to race and health literacy. Health Educ Res. 2013 Jun;28(3):502-11. doi: 10.1093/her/cyt043. Epub 2013 Mar 22. PMID 23525779
- [Result] Allen KD, Oddone EZ, Stock JL, Coffman CJ, Lindquist JH, Juntilla KA, Lemmerman DS, Datta SK, Harrelson ML, Weinberger M, Bosworth HB. The Self-Management of OsteoArthritis in Veterans (SeMOA) Study: design and methodology. Contemp Clin Trials. 2008 Jul;29(4):596-607. doi: 10.1016/j.cct.2007.11.004. Epub 2007 Nov 22. PMID 18206425
- [Result] Allen KD, Oddone EZ, Coffman CJ, Keefe FJ, Lindquist JH, Bosworth HB. Racial differences in osteoarthritis pain and function: potential explanatory factors. Osteoarthritis Cartilage. 2010 Feb;18(2):160-7. doi: 10.1016/j.joca.2009.09.010. Epub 2009 Oct 1. PMID 19825498
- [Result] Allen KD, Oddone EZ, Coffman CJ, Datta SK, Juntilla KA, Lindquist JH, Walker TA, Weinberger M, Bosworth HB. Telephone-based self-management of osteoarthritis: A randomized trial. Ann Intern Med. 2010 Nov 2;153(9):570-9. doi: 10.7326/0003-4819-153-9-201011020-00006. PMID 21041576
- See also: Durham VA HSR&D Center of Excellence (Study Site) — http://www.durham.hsrd.research.va.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on Oct 3, 2006 and ended on June 30, 2008. We used VA medical records to identify patients with hip and knee OA and no exclusionary diagnoses. We mailed introductory letters to these individuals and followed up with a screening phone call. Eligible patients were asked to come to the Durham VA for a baseline visit.
Groups:
- Arm 1: Health Education Intervention
  Health Education: 12-month intervention consisting of monthly phone calls about common health conditions and screening. Also includes written educational materials on these topics.
- Arm 2: Usual Medical Care
- Arm 3: Osteoarthritis Self-Management
  Osteoarthritis Self-Management: 12-month intervention consisting of monthly phone calls about topics related to self-care for osteoarthritis. Also includes written educational materials on these topics. Participants set goals and action plans, with assistance from health educator, about managing their osteoarthritis.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3
Started | 175 | 174 | 174
Completed | 158 | 157 | 146
Not Completed | 17 | 17 | 28
Not completed — Developed exclusion criterion | 4 | 6 | 7
Not completed — Lost to Follow-up | 9 | 6 | 9
Not completed — Withdrawal by Subject | 4 | 5 | 12

BASELINE CHARACTERISTICS:
Population: Among n=523 who consented and were randomized 8 were excluded from analyses because subsequent review of VA medical records revealed there was no documentation of radiographic evidence of knee or hip OA and therefore these participants did not meet initial eligibility requirements.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Total
Number analyzed (Participants) | 172 | 171 | 172 | 515
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (10.8) | 59.7 (10.1) | 60.3 (10.3) | 60.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 15 | 37
  Male | 160 | 161 | 157 | 478
Race/Ethnicity, Customized [Number; unit: participants]
  White | 91 | 92 | 95 | 278
  Non-White | 81 | 79 | 77 | 237
Region of Enrollment [Number; unit: participants]
  United States | 172 | 171 | 172 | 515

OUTCOME MEASURES:

1. Primary Outcome: Pain
Description: Arthritis Impact Measurement Scales-2 (AIMS2), which consists of five items assessing typical pain, pain severity, and pain during specific times of the day, using a 5-point Likert scale ("all days" to "no days"). The possible range of scores is 0-10, with higher scores indicating more severe pain.
Time Frame: Baseline and 12-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 172 | 171 | 172
units on a scale
  Baseline | 6.01 (2.28) | 5.77 (2.14) | 5.92 (2.27)
  12-Month Follow-Up | 5.84 (2.32) | 5.46 (2.03) | 5.22 (2.44)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 3; Primary hypothesis: OA self-management intervention results in greater improvement in AIMS2 pain score than usual care or health education control. Sample size estimate based on detecting 0.57 point (14%) difference between groups. Analyses were linear mixed models, intent-to-treat basis; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.0 to 0.2] — The mean difference (final values) is based on differences in the outcome between study groups at 12-month follow-up, in the context of the mixed models
Statistical Analysis 2: Comparison: Arm 2 vs Arm 3; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.105, Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.8 to 0.1] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: AIMS 2 Physical Function
Description: The AIMS2 physical function subscale includes 28 items that measure aspects of mobility, walking and bending, hand and finger function, arm function, self-care, and household tasks. All items on the AIMS2 physical function subscale are measured on a 5-point Likert scale ("all days" to "no days"). Scores can range from 0-10, with higher scores indicating worse function.
Time Frame: Baseline and 12-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 172 | 171 | 172
units on a scale
  Baseline | 2.70 (1.78) | 2.27 (1.34) | 2.60 (1.68)
  12-Month Follow-Up | 2.87 (1.94) | 2.34 (1.55) | 2.57 (1.77)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 3; Secondary hypothesis: OA self-management intervention results in greater improvement in AIMS2 function score than usual care or health education control. Analyses were linear mixed models, intent-to-treat basis; Test type: Superiority or Other; p = 0.093, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm 2 vs Arm 3; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.43, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to 0.2] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: AIMS 2 Affect
Description: The AIMS2 affect subscale includes ten items that encompass mood and tension. All items on the AIMS2 affect subscale are measured on a 5-point Likert scale ("all days" to "no days"). Scores can range from 0-10, with higher scores indicating worse affect.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 172 | 171 | 172
units on a scale
  Baseline | 3.64 (2.26) | 3.23 (2.04) | 3.74 (2.29)
  12-Month Follow-Up | 3.44 (2.20) | 3.08 (2.09) | 3.58 (3.35)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 3; Secondary hypothesis: OA self-management intervention results in greater improvement in AIMS2 affect score than usual care or health education control. Analyses were linear mixed models, intent-to-treat basis; Test type: Superiority or Other; p = 0.78, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.3 to 0.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm 2 vs Arm 3; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.79, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.3 to 0.4] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Arthritis Self Efficacy
Description: The Arthritis Self-Efficacy Scale measures how certain patients are they can perform 8 specific activities or tasks, related to arthritis. Items are scored on a Likert Scale (1=very uncertain to 10=very certain), with total scores ranging from 1-10. Higher scores indicate greater arthritis self-efficacy.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 172 | 171 | 172
units on a scale
  Baseline | 5.78 (2.01) | 5.92 (1.92) | 5.68 (2.07)
  12-Month Follow-Up | 5.80 (2.06) | 5.96 (1.96) | 6.09 (2.13)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 3; Secondary hypothesis: OA self-management intervention results in greater improvement in arthritis self-efficacy score than usual care or health education control. Analyses were linear mixed models, intent-to-treat basis; Test type: Superiority or Other; p = 0.043, Mixed Models Analysis; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [0.0 to 0.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm 2 vs Arm 3; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.066, Mixed Models Analysis; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [0.0 to 0.7] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Description: We have entered adverse events in relatively broad categories (e.g., Hospital Admission, Emergency Room Visit) because this was what was collected in order to meet reporting requirements of the IRB. More specific adverse event data was not required or collected, and none of the adverse events were study related.
Arm/Group | Arm 1 | Arm 2 | Arm 3
Serious Adverse Events (participants affected / at risk) | 10/175 | 7/174 | 14/174
Other Adverse Events (participants affected / at risk) | 33/175 | 25/174 | 36/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=175) | Arm 2 (N=174) | Arm 3 (N=174)
Death (General disorders) | 0 | 0 | 1 — Not Study Related
Hospital Admission (Cardiac disorders) | 2 | 3 | 7 — Not Study Related
Hospital Admission (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 — Not Study Related
Hospital Admission (Infections and infestations) | 0 | 0 | 1 — Not Study Related
Hospital Admission (General disorders) | 0 | 0 | 1 — Not Study Related
Inpatient Surgery (Surgical and medical procedures) | 4 | 6 | 7 — Not Study Related
Significant Disability (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 — Not Study Related
Hospital Admission (Renal and urinary disorders) | 1 | 1 | 0 — Not Study Related
Hospital Admission (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — Not Study Related
Hospital Admission (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 — Not Study Related
Hospital Admission (Endocrine disorders) | 1 | 0 | 0 — Not Study Related
Significant Disability (Nervous system disorders) | 1 | 0 | 0 — Not Study Related
Hospital Admission (Hepatobiliary disorders) | 0 | 1 | 0 — Not Study Related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=175) | Arm 2 (N=174) | Arm 3 (N=174)
Emergency Room Visit (Gastrointestinal disorders) | 2 | 0 | 6 — Not study-related
Emergency Room Visit (Musculoskeletal and connective tissue disorders) | 20 | 7 | 19 — Not study related
Emergency Room Visit (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 7 — Not study related
Emergency Room Visit (General disorders) | 11 | 11 | 13
Emergency Room Visit (Cardiac disorders) | 0 | 0 | 2 — Not Study Related
Emergency Room Visit (Ear and labyrinth disorders) | 0 | 0 | 1 — Not Study Related
Emergency Room Visit (Renal and urinary disorders) | 1 | 1 | 1 — Not Study Related
Outpatient Surgery (Surgical and medical procedures) | 10 | 10 | 14 — Not Study Related
Emergency Room Visit (Psychiatric disorders) | 2 | 1 | 0 — Not Study Related
Emergency Room Visit (Vascular disorders) | 1 | 0 | 0 — Not Study Related
Emergency Room Visit (Eye disorders) | 1 | 1 | 0 — Not Study Related
Emergency Room Visit (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 — Not Study Related
Emergency Room Visit (Infections and infestations) | 1 | 0 | 0 — Not Study Related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes